CLINICAL TRIAL: NCT04944381
Title: a Voluntary, Investigator-initiated, Inactivated COVID-19 Vaccine Controlled Clinical Trial of COVID-19 mRNA Vaccine in Adults Aged 18 Years and Above
Brief Title: Study of Ameliorating Effect of COVID-19 mRNA Vaccine in Individuals Immunized With Inactivated Vaccine
Acronym: COVID-19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Qihan Li (Unknown)
Responsible Party: Sponsor-Investigator, Qihan Li, Director, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20210624
Record Dates: First submitted 2021-06-24; First posted 2021-06-29 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: SARS-CoV-2 Acute Respiratory Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SARS-Cov-2 mRNA vaccine immunization group (Experimental): The 98 participants will be inoculated with one dose SARS-Cov-2 mRNA vaccine from Stemirna Therapeutics Co., Ltd.
  Interventions: Biological: SARS-Cov-2 mRNA vaccine immunization
- Inactivated SARS-Cov-2 vaccine immunization group (Experimental): The 14 participants will be inoculated with one dose inactivated SARS-Cov-2 vaccine from institute of medical biology, Chinese academy of medical sciences(IMBCAMS).
  Interventions: Biological: Inactivated SARS-Cov-2 vaccine immunization

INTERVENTIONS:
Biological: SARS-Cov-2 mRNA vaccine immunization — The 98 participants will be inoculated with one dose SARS-Cov-2 mRNA vaccine from Stemirna Therapeutics Co., Ltd and .
  Arms: SARS-Cov-2 mRNA vaccine immunization group
Biological: Inactivated SARS-Cov-2 vaccine immunization — The 14 participants will be inoculated with one dose inactivated SARS-Cov-2 vaccine from institute of medical biology, Chinese academy of medical sciences(IMBCAMS).
  Arms: Inactivated SARS-Cov-2 vaccine immunization group

SUMMARY:
this is a voluntary, investigator-initiated, inactivated COVID-19 vaccine controlled clinical trial to evaluate the immunogenicity and safety of COVID-19 mRNA vaccine in adults aged 18 years and above which have immunized with two dose of inactivated COVID-19 vaccine at least 6 months ago.

DETAILED DESCRIPTION:
A total of 112 participants will be enrolled in the study. All the participants have immunized with two doses of inactivated COVID-19 vaccine at least 6 months ago. The 98 participants will be inoculated with one dose COVID-19 messenger ribonucleic acid(mRNA) vaccine from Stemirna Therapeutics Co., Ltd and the others will be inoculated with one dose inactivated COVID-19 vaccine from institute of medical biology, Chinese academy of medical sciences(IMBCAMS). Before the inoculation, 14 days and 28 days after the immunization, blood samples will be taken for determination of neutralizing antibody and immunoglobulin G(IgG) antibody against severe acute respiratory syndrome coronavirus 2(SARS-CoV-2) N protein and S protein (enzyme-linked immuno sorbent assay, ELISA method); and before the inoculation and 28 days after the immunization, blood samples will be taken for detecting specific T cells with the enzyme-linked immunospot(ELISPOT) assay with an aim to evaluate immunogenicity. Safety observations for all participants will be conducted from the inoculation to 28 days, and follow-up of severe adverse events (SAEs) will also be conducted from inoculation to at least 12 months to evaluate the safety of the investigational vaccine.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 years and above (including boundary values), both female and male.
2. Legal identification of the participants shall be provided.
3. the participants have inoculation two doses of inactivated SARS-CoV-2 vaccine (vero cell) was manufactured by IMBCAMS at least 6 months ago.
4. Participants shall understand the content in the Informed Consent Form (ICF) and the vaccine for administration, sign the ICF voluntarily and are capable of using thermometers and rulers, and filling in diary cards and contact cards as per the requirements.
5. Subject shall be able to communicate well with investigators, understand and comply with the requirements of this study.
6. Participants with oral temperature ≤ 37.9 ℃.
7. Female participants of childbearing potential (defined as any female who has experienced menarche and who is NOT surgically sterile [i.e., hysterectomy, bilateral tubal ligation, or bilateral oophorectomy] or postmenopausal [defined as amenorrhea at least 12 consecutive months]) must agree to be heterosexually inactive OR consistently use any of the following methods of contraception: a) Condoms (male or female) b) Diaphragm with spermicide c) Cervical cap with spermicide d) Intrauterine device e) Oral or patch contraceptives f) Any country regulatory-approved contraceptive method that is designed to protect against pregnancy g) Abstinence, as a form of contraception, is acceptable if in line with the participant's lifestyle (other approaches to abstinence are not acceptable).

Exclusion Criteria:

1. Contraindications to commonly used vaccines;
2. History of allergy to any vaccines or drug;
3. Received any vaccine within 1 month before the vaccination；
4. Serious diseases required to be excluded, including but not limited to history of diseases in nervous system, cardiovascular system, blood and lymphatic system, immune system, kidney, liver, gastrointestinal tract, respiratory system, metabolism, bones and other systems, and a history of malignant tumors;
5. Before immunizing the investigational vaccine, those who developed acute disease within 2 weeks, or had symptoms of fever or upper respiratory tract infection within 7 days;
6. Those who have a hereditary bleeding tendency or blood coagulation dysfunction, or a history of thrombosis or hemorrhagic disease；
7. Surgical removal of whole or part of spleen for any reason；
8. Those who have undergone surgery within 3 months before signing the ICF or those who plan to undergo surgery during or within 3 months after completion of the trial (including plastic surgery, dental and oral surgery);
9. Those who donated or lost blood (≥400 mL) in the past 3 months, who received blood transfusion or use of blood products, or who plan blood donation during the trial;
10. Those who received other investigational or unregistered products (drugs, vaccines, biological product or devices) in the past 3 months before signing the ICF, or plan to use them during the study.
11. Those who received immunosuppressant therapy within 6 months before signing the ICF, such as long-term systemic glucocorticoid treatment (with systemic glucocorticoid therapy for more than 2 consecutive weeks within 6 months, such as prednisone or similar drugs), but local administration is permitted (such as ointment, eye drops, inhalants, or nasal spray). The local administration should not exceed the recommended dose in the package insert or have any signs of systemic exposure;
12. Participants cannot meet the criteria through the comprehensive physical examination, mainly including: - Abnormal vital signs with clinical significance (awakening heart rate <55 beats/min or >100 beats/min, systolic blood pressure ≥140 millimetre of mercury (mmHg) or diastolic blood pressure ≥90mmHg); - Those who tested positive for type 1 or type 2 human immunodeficiency virus (HIV-1/2) antibody, or SARS-CoV-2 nucleic acid;
13. History of COVID-19;
14. Participants who have a positive pregnancy test, or are breastfeeding, or planning pregnancy, or plan to donate sperm or eggs within 12 months from the screening period to the whole-course immunization;
15. Participants who are considered as inappropriate for the trial by investigators.
16. Suspected or known current alcohol or drug dependency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2021-07-02 (Estimated); Primary Completion 2021-08-02 (Estimated); Study Completion 2022-08-02 (Estimated)

PRIMARY OUTCOMES:
the geometric mean titer (GMT) of neutralizing antibody | 14 days and 28 days
  the geometric mean titer (GMT) of neutralizing antibody against SARS-Cov-2 14 days and 28 days after vaccine inoculation
the incident of solicited adverse events(AEs) | 7 days
  the incident of solicited AEs at the inoculation (local) and solicited AEs at the non-inoculation (systemic) within 7 days after immunization.

SECONDARY OUTCOMES:
The Geometric Mean Titer (GMT) of IgG antibody | 14 days and 28 days
  The Geometric Mean Titer (GMT) of IgG antibody against SARS-CoV-2 N protein and S protein (ELISA method) 14 days and 28 days after vaccine inoculation
Specific T cells with ELISPOT assay | 28 days
  Detecting specific T cells with ELISPOT assay 28 days after vaccine inoculation
The incidence of AEs | 28 days
  The incidence of AEs from the inoculation to 28 days after the immunization.
The incidence of SAEs | 1 year
  The incidence of AEs from the inoculation to at least 12 months after the immunization.

IPD SHARING:
Plan to Share IPD: No